CLINICAL TRIAL: NCT01631227
Title: A Prospective, Randomized Double-blind Parallel Group Study to Compare the Effect of Eprosartan and Eprosartan Mesylate on Blood Pressure in Subjects With Mild to Moderate Essential Hypertension
Brief Title: Comparison of the Effect of Eprosartan and Eprosartan Mesylate on Blood Pressure in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Quintiles, Inc. (Industry); Synexus (Other); author! et al. BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-385; 2010-019432-12 (EudraCT Number)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — eprosartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eprosartan (Experimental): Eprosartan + Placebo Eprosartan Mesylate
  Interventions: Drug: Eprosartan; Drug: Placebo Eprosartan mesylate
- Eprosartan Mesylate (Active Comparator): Eprosartan Mesylate + Placebo Eprosartan
  Interventions: Drug: Eprosartan Mesylate; Drug: Placebo Eprosartan

INTERVENTIONS:
Drug: Eprosartan — Eprosartan 450 mg
  Arms: Eprosartan
Drug: Eprosartan Mesylate — Eprosartan mesylate 600 mg
  Other Names: ABT-139; Teveten
  Arms: Eprosartan Mesylate
Drug: Placebo Eprosartan mesylate — Placebo Eprosartan mesylate
  Other Names: Placebo
  Arms: Eprosartan
Drug: Placebo Eprosartan — Placebo Eprosartan
  Other Names: Placebo
  Arms: Eprosartan Mesylate

SUMMARY:
Aim of this study is to compare the blood pressure lowering effect of a new drug formulation of eprosartan. Eprosartan belongs to a class of blood pressure lowering agents used worldwide since years with proven efficacy. The new formulation is compared to the currently marketed eprosartan tablet. Equivalent efficacy in blood pressure lowering effects should be demonstrated.

ELIGIBILITY:
Inclusion Criteria

* Males or females with essential hypertension, blood pressure values between 140 mmHg and 179 mmHg systolic and between 90 mmHg and 109 mmHg diastolic
* Given written informed consent prior to starting the study

Exclusion Criteria

* Women with childbearing potential, breast feeding or pregnant;
* Inability to discontinue all prior antihypertensive medication;
* Secondary hypertension
* Severe hypertension
* Severe diabetes mellitus (HbA1c greater 8.5%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri N. Kazei, MD, Study Director — Abbott Healthcare Products B.V.
Locations (38):
- Germany (13):
  - Site Reference ID/Investigator# 74062, Berlin
  - Site Reference ID/Investigator# 74066, Bochum
  - Site Reference ID/Investigator# 74065, Dresden
  - Site Reference ID/Investigator# 93513, Dresden
  - Site Reference ID/Investigator# 93495, Essen
  - Site Reference ID/Investigator# 93515, Frankfurt
  - Site Reference ID/Investigator# 74060, Frankfurt
  - Site Reference ID/Investigator# 74063, Görlitz
  - Site Reference ID/Investigator# 93494, Hamburg
  - Site Reference ID/Investigator# 93493, Karlsruhe
  - Site Reference ID/Investigator# 74061, Leipzig
  - Site Reference ID/Investigator# 74064, Magdeburg
  - Site Reference ID/Investigator# 93514, Nuremberg
- Russia (15):
  - Site reference ID/Investigator # 82515, Barnaul
  - Site reference ID/Investigator # 82520, Kazan'
  - Site reference ID/Investigator # 82493, Kemerovo
  - Site reference ID/Investigator # 82516, Kemerovo
  - Site refernce ID/Investigator # 82521, Krasnodar
  - Site reference ID/Investigator # 82495, Novosibirsk
  - Site reference ID/Investigator # 82494, Novosibirsk
  - Site reference ID/Investigator # 82525, Novosibirsk
  - Site reference ID/Investigator # 82522, Saint Petersburg
  - Site reference ID/Investigator # 82517, Saint Petersburg
  - Site reference ID/Investigator # 82524, Saint Petersburg
  - Site reference ID/Investiragor # 82523, Saint Petersburg
  - Site reference ID/Investigator # 82519, Saint Petersburg
  - Site reference ID/Investigator # 82518, Saint Petersburg
  - Site reference ID/Investigator # 82527, Saint Petersburg
- United Kingdom (10):
  - Site Reference ID/Investigator# 74057, Birmingham
  - Site Reference ID/Investigator# 74059, Cardiff
  - Site Reference ID/Investigator# 74056, Chorley
  - Site Reference ID/Investigator# 74054, Glasgow
  - Site reference ID/Investigator # 95456, Glasgow
  - Site Reference ID/Investigator# 74053, Liverpool
  - Site reference ID/Investigator # 95457, London
  - Site Reference ID/Investigator# 74055, Manchester
  - Site reference ID/Investigator # 95455, Northwood
  - Site Reference ID/Investigator# 74058, Reading

RESULTS

PARTICIPANT FLOW:
Groups:
- Eprosartan: Eprosartan 450 mg + Placebo Eprosartan Mesylate
- Eprosartan Mesylate: Eprosartan Mesylate 600 mg + Placebo Eprosartan
Period: Overall Study
Arm/Group | Eprosartan | Eprosartan Mesylate
Started | 333 | 332
Safety Subject Sample | 332 (1 patient was randomized by mistake and never received study medication.) | 332
Full Analysis Set Population | 330 (2 patients not eligible for the Full Analysis Set due to missing post-baseline efficacy measurement) | 331 (1 patient not eligible for the Full Analysis Set due to missing post-baseline efficacy measurement)
Completed | 303 | 310
Not Completed | 30 | 22
Not completed — withdrawn consent | 27 | 21
Not completed — Adverse Event | 1 | 0
Not completed — administrative | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set consists of 330 and 331 patients respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eprosartan | Eprosartan Mesylate | Total
Number analyzed (Participants) | 333 | 332 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 60 (10) | 60 (10)
Gender [Number; unit: participants]
  Female | 186 | 201 | 387
  Male | 144 | 130 | 274

OUTCOME MEASURES:

1. Primary Outcome: Assess the Therapeutic Equivalence of Eprosartan (a New Formulation Containing Only the Active Moiety Eprosartan) With Eprosartan Mesylate (Currently Marketed Formulation) on Change of Sitting Diastolic Blood Pressure (DBP) From Baseline
Description: Change from baseline of diastolic blood pressure (DBP), sitting
Time Frame: 8 weeks
Population: Full analysis subject sample
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Eprosartan | Eprosartan Mesylate
Number analyzed (Participants) | 330 | 331
mmHg | -7.4 (7.7) | -7.2 (7.5)

ADVERSE EVENTS:
Time Frame: 15 weeks (3 run-in and 12 weeks treatment)
Arm/Group | Eprosartan | Eprosartan Mesylate
Serious Adverse Events (participants affected / at risk) | 3/332 | 7/332
Other Adverse Events (participants affected / at risk) | 15/332 | 18/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eprosartan (N=332) | Eprosartan Mesylate (N=332)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
THYROID CYST (Endocrine disorders) | 0 (0) | 1 (1)
CYSTIC RUPTURE (General disorders) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MENISCAL DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eprosartan (N=332) | Eprosartan Mesylate (N=332)
NASOPHARYNGITIS (Infections and infestations) | 15 (15) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less